CLINICAL TRIAL: NCT04382560
Title: Resting Heart Rate Variability as a Predictor of Coping Strategies and Responsiveness to a Brief Online Intervention During Forced Quarantine
Brief Title: Coping Strategies and Responsiveness to a Brief Online Intervention During COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: University of Roma La Sapienza (Other); King's College London (Other)
Responsible Party: Principal Investigator, Luca Carnevali, PhD, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ESPCOV1
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Behavior, Social; Autonomic Imbalance
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Intervention Model Description: wait-list control design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a Deep Breathing Training and a Compassion Intervention. Deep Breathing Training and Compassion Intervention will be administered once, on two consecutive days, and will last for 30 minutes.
  Interventions: Other: Deep Breathing training; Other: Compassion focused intervention
- Wait-list control group (No Intervention): The waiting list group will receive the intervention at the end of the study.

INTERVENTIONS:
Other: Deep Breathing training — The intervention will comprise a psychoeducational part on the theorethical background underlying this technique and a pratical session in which partecipant will be instructed to inhale air with his/her nose and exhale with his/her mouth for a period of 3 seconds of inhalation and 7 seconds of exhalation (i.e., 6 cycles of breaths per minute;). During the session, the participant will be encouraged to put one hand over his/her chest and the other over the abdomen in order to see the difference between normal breathing and deep breathing. To help the subjects in the training, an online pacer will give the rhythm of respiration and will be used as visual feedback.
  Arms: Intervention group
Other: Compassion focused intervention — The short compassion focused intervention will begin with a short psychoeducation on the evolved nature and difficulties of the human mind, such as tendencies for negativity bias, negative rumination, and self-criticism. Participants will then be offered insights into how humans can work with their 'tricky brains' using body-based and psychological-based practices aimed at increasing a grounding and soothing compassionate attitude towards ourselves and others. In particular, participants will be instructed to pratice a mindfulness technique designed to help them to become more aware of their present moment-to-moment and more compassionate towards their own emotions. They will then be guided to create an image conveying warmth and compassion to them. Lastly, participants will be guided to bring the image to mind and then write write a brief "self-compassionate letter" to themselves from that point of view.
  Arms: Intervention group

SUMMARY:
The present study investigates the efficacy of a brief and cost-effective video-intervention that combines bottom-up elements of deep breathing and third-wave cognitive behavioral therapy techniques (i.e., mindfulness and compassion) on coping strategies during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Previous participation (maximum elapsed time: 2.0 years) in a study conducted by the same research group and incorporating cardiac autonomic assessment at rest

Exclusion Criteria:

* Self-reported development of cardiovascular disease since previous assessment
* Use of psychotropic medications or medications affecting the autonomic nervous system

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Dispositional questionnaire 1 | During waking hours for two consecutive days before the intervention/control condition
  Perseverative cognition measured as frequency score. Minimum score = 0 Maximum score = 28. Higher scores mean a worse outcome.
Dispositional questionnaire 1 | During waking hours for two consecutive days after the intervention/control condition
  Perseverative cognition measured as frequency score. Minimum score = 0 Maximum score = 28. Higher scores mean a worse outcome.
Dispositional questionnaire 2 | During waking hours for two consecutive days after the intervention/control condition
  Effective coping strategies measured as frequency score. Minimum score = 0 Maximum score = 28. Higher scores mean a better outcome.
Dispositional questionnaire 3 | During waking hours for two consecutive days before the intervention/control condition
  Mood state measured as score on a Likert scale. Minimum score = 1 Maximum score = 5. Higher scores mean a worse outcome.
Dispositional questionnaire 3 | During waking hours for two consecutive days after the intervention/control condition
  Mood state measured as score on a Likert scale. Minimum score = 1 Maximum score = 5. Higher scores mean a worse outcome.
Dispositional questionnaire 4 | During waking hours for two consecutive days before the intervention/control condition
  Emotional state measured as score on a Likert scale. Minimum score = 1 Maximum score = 5. Higher scores mean a worse outcome.
Dispositional questionnaire 4 | During waking hours for two consecutive days after the intervention/control condition
  Emotional state measured as score on a Likert scale. Minimum score = 1 Maximum score = 5. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Heart rate | During waking hours for two consecutive days before the intervention/control condition
  Heart rate (measured in beats per minute) recorded via a smartphone application
Heart rate | During waking hours for two consecutive days after the intervention/control condition
  Heart rate (measured in beats per minute) recorded via a smartphone application
Cardiac vagal modulation | During waking hours for two consecutive days before the intervention/control condition
  Root mean square of the successive differences (measured in ms) recorded via a smartphone application
Cardiac vagal modulation | During waking hours for two consecutive days after the intervention/control condition
  Root mean square of the successive differences (measured in ms) recorded via a smartphone application

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No